CLINICAL TRIAL: NCT00228553
Title: A 12-Month, Open-Label, Flexible-Dosage (100 to 250 mg/Day) Extension Study of the Safety and Efficacy of Armodafinil (CEP-10953) in the Treatment of Patients With Excessive Sleepiness Associated With Narcolepsy, Obstructive Sleep Apnea/Hypopnea Syndrome, or Chronic Shift Work Sleep Disorder (With an Open-Ended Extension Period)
Brief Title: Extension Study of the Safety and Efficacy of Armodafinil in the Treatment of Patients With Excessive Sleepiness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C10953/3024/ES/MN
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Excessive Daytime Sleepiness; Narcolepsy; Obstructive Sleep Apnea/Hypopnea Syndrome; Chronic Shift Work Sleep Disorder
MeSH Terms: conditions — Disorders of Excessive Somnolence; Narcolepsy; Sleep Apnea, Obstructive

ARMS (1):
- 1 (Experimental): Armodafinil 100 to 250 mg/day
  Interventions: Drug: Armodafinil 100 to 250 mg/day

INTERVENTIONS:
Drug: Armodafinil 100 to 250 mg/day — Armodafinil 100-250 mg: once daily in the morning for patients with obstructive sleep apnea/hypopnea syndrome (OSAHS) or narcolepsy, once daily only on nights worked for patients with shift worker sleep disorder (SWSD).

SUMMARY:
A 12 Month, Open-Label, Flexible Dosage Extension Study of the Safety and Efficacy of Armodafinil (CEP-10953) in the Treatment of Patients with Excessive Sleepiness Associated with Narcolepsy, Obstructive Sleep Apnea/Hypopnea Syndrome, or Chronic Shift Work Sleep Disorder

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* Men and women (outpatients) of any ethnic origin, between 18 and 65 years of age (inclusive) at the beginning of the respective double-blind study, are eligible.
* The patient has completed a cephalon-sponsored double-blind study (study C10953/3020/NA/MN, C10953/3021/AP/MN, C10953/3022/CM/MN, or C10953/3025/AP/MN), and the investigator has recommended they be enrolled.
* Patients with OSAHS must continue to be regular users of nCPAP therapy, which the investigator considers to remain effective. Patients with chronic SWSD must work 5 nights/month, with night shifts including at least 6 hours between 2200 and 0800 that are no longer than 12 hours in duration.
* The patient is considered to be in good health.
* Women must be surgically sterile, 2 years postmenopausal, or if of childbearing potential, must use a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, implanted, and Depo-Provera contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]).
* The patient must be willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* Have any clinically significant, uncontrolled medical conditions (treated or untreated).
* Have a probable diagnosis of a current sleep disorder other than the primary diagnosis of narcolepsy, OSAHS, or chronic SWSD.
* Consume caffeine including coffee, tea and/or other caffeine-containing beverages or food averaging more than 600 mg of caffeine.
* Use any prescription drugs disallowed by the protocol or clinically significant use of over-the-counter (OTC) drugs within 7 days before visit 1.
* Have a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM-IV) (American Psychiatric Association 1994).
* Have a positive urine drug screen (UDS) (subjects enrolling in this open-label study within 7 days after completing the double-blind study may be enrolled without UDS results).
* Have a clinically significant deviation from normal in the physical examination.
* Are pregnant or lactating. Any woman becoming pregnant during the study will be withdrawn from the study.
* Have any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* Have a known clinically significant drug sensitivity to stimulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2004-05; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Director, MD, Study Director — Cephalon
Locations (100):
- United States (74):
  - Sleep Disorders Ctr of Alabama, Birmingham, Alabama
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Psypharma Clinical Research, Phoenix, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Advanced Clinical Research Ins, Anaheim, California
  - Southwestern Research, Beverly Hills, California
  - Pacific Sleep Medicine Service, Los Angeles, California
  - Pacific Sleep Medicine Service, Palm Springs, California
  - Radiant Research San Diego, San Diego, California
  - Pacific Sleep Medicine Service, San Diego, California
  - BMR HealthQuest, San Diego, California
  - Sleep Clinic of San Francisco, San Francisco, California
  - St. Johns Medical Plaza Sleep, Santa Monica, California
  - Stanford University, Stanford, California
  - PAB Clinical Research, Brandon, Florida
  - St. Petersburg Sleep Disorder, St. Petersburg, Florida
  - Sleep-Wake Disorder Center, Winter Park, Florida
  - Neurotrials Research, Atlanta, Georgia
  - Sleep Disorders Center of GA, Atlanta, Georgia
  - SLEEPMED, Inc., Macon, Georgia
  - Radiant Research Marietta, Marietta, Georgia
  - Henry Lahmeyer, MD, Northfield, Illinois
  - Peoria Pulmonary Associates, Peoria, Illinois
  - Center for Sleep Disorders, Danville, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - Vince and Associates Clinical, Overland Park, Kansas
  - Topeka Pulmonary, Topeka, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Community Research, Crestview, Kentucky
  - Chest Medicine Associates DBA, Louisville, Kentucky
  - Neurotrials Research of New Or, Metairie, Louisiana
  - Northshore Research Associates, Slidell, Louisiana
  - Center for Sleep/Wake Disorder, Chevy Chase, Maryland
  - Regional Pulmonary and Sleep, Elkton, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - Sleep Disorders Center, Hattiesburg, Mississippi
  - Washington University School o, St Louis, Missouri
  - Clinical Rsch Center of Nevada, Las Vegas, Nevada
  - CNS Research Institute, Clementon, New Jersey
  - New York University, New York, New York
  - Clinilabs / Sleep Disorders In, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - Vital re:Search, Greensboro, North Carolina
  - Neurology Associates of Hickor, Hickory, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Central Carolina Neurology Sle, Salisbury, North Carolina
  - All Trials Clinical Research, Winston-Salem, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - North Coast Clinical Trials, Beechwood, Ohio
  - Community Research Management, Cincinnati, Ohio
  - Tri State Sleep Disorders Cent, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dept Veterans Affairs Dayton, Dayton, Ohio
  - Ohio Sleep Medicine-Neurosci, Dublin, Ohio
  - Southwest Cleveland Sleep Cent, Middleburg Heights, Ohio
  - St. Vincent Mercy Medical Cent, Toledo, Ohio
  - Clinical Pharmaceutical Trials, Tulsa, Oklahoma
  - Capital Region Sleep Disorders, Carlisle, Pennsylvania
  - Consolidated Clinical Trials, Pittsburgh, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Lowcountry Lung and Critical, Charleston, South Carolina
  - SleepMed of South Carolina, Columbia, South Carolina
  - St. Thomas Sleep Disorders Cen, Nashville, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Sleep Medicine Institute, Dallas, Texas
  - Houston Sleep Center, Houston, Texas
  - VA Medical CenterSleep Diagnos, Houston, Texas
  - Sadler Clinic, The Woodlands, Texas
  - Radiant Research Salt Lake, Salt Lake City, Utah
  - Sentara Norfolk General Hospit, Norfolk, Virginia
  - Swedish Sleep Medicine Institute, Seattle, Washington
  - Allegiance Research Specialist, Wauwatosa, Wisconsin
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Monash Medical Center, Clayton, Victoria
  - Melbourne Sleep Disorders Ctr., East Melbourne, Victoria
- Canada (8):
  - Canadian Sleep Institute, Calgary, Alberta
  - Sleep Clinic, Kitchener, Ontario
  - Niagara Clinical Research, Niagara Falls, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - West Parry Sound Health Center, Parry Sound, Ontario
  - Sleep and Neuropsychiatry Cent, Scarborough Village, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Baycrest Hospital, Toronto, Ontario
- France (4):
  - Hopital Guy de Chauliac, Montpellier, Cedex 05
  - Universitaires de Strasbourg, Strasbourg, Cedex
  - Hopital Antoine Beclere, Clamart, Clamart
  - Hospital Henri-Mondor, Créteil
- Germany (4):
  - University of Freiburg, Freiburg im Breisgau
  - Klinikum der Philipps, Marburg
  - University of Regensburg, Regensburg
  - Hephata Klinik, Schwalmstadt
- SomniCare Sleep Institute, San Juan, Puerto Rico
- Russia (4):
  - City Clinical Hospital 33, Moscow
  - City Clinical Hospital 83, Moscow
  - Clinical Hospital Russian Scie, Saint Petersburg
  - Multifunction Center of Neurol, Samara

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 99 centers in the US, Canada, France, Germany, Russia, and Australia. First participant enrolled: 15 May 2004/ Last participant last visit: 19 July 2006
Pre-assignment Details: 12 participants (3 female ; 9 male) withdrew after randomization but prior to receiving study drug
Period: Overall Study
Arm/Group | Armodafinil 100 to 250 mg/Day
Started | 743
Completed | 313
Not Completed | 430
Not completed — Adverse Event | 112
Not completed — Lack of Efficacy | 34
Not completed — Lost to Follow-up | 67
Not completed — Physician Decision | 48
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 115
Not completed — Pregnancy | 2
Not completed — Miscellaneous | 46

BASELINE CHARACTERISTICS:
Arm/Group | Armodafinil 100 to 250 mg/Day
Number analyzed (Participants) | 731
Age, Categorical [Count of Participants; unit: Participants] — 12 participants (3 female ; 9 male) withdrew after randomization but prior to receiving study drug
  Participants
    <=18 years | 0
    Between 18 and 65 years | 726
    >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants] — 12 participants (3 female ; 9 male) withdrew after randomization but prior to receiving study drug
  Participants
    Female | 257
    Male | 474
Region of Enrollment [Number; unit: participants]
  France | 8
  United States | 611
  Canada | 70
  Australia | 25
  Russian Federation | 16
  Germany | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability in This Patient Population (Narcolepsy, OSAHS, SWSD) Over Time (up to 2 Years)
Description: An adverse event is any untoward medical occurrence in a patient that develops or worsens in severity during the conduct of a clinical study. Serious and Non-serious Adverse Events (SAEs). Serious adverse event is any adverse event occurring at any dose that results in any of the following outcomes: death, life-threatening, inpatient hospitalization, persistent or significant disability, congenital anomaly, or an important medical event. An adverse event that does not meet any of the criteria for seriousness listed previously will be regarded as a nonserious adverse event.
Time Frame: End of months 1, 3, 6, 9, and 12 and every 3 months for up to an additional year
Population: Safety Analysis set of 731 total patients: 12 participants (3 female ; 9 male) withdrew after randomization but prior to receiving study drug.
Measure: Number; unit: Participants
Arm/Group | Armodafinil 100 to 250 mg/Day
Number analyzed (Participants) | 731
Participants | 667

ADVERSE EVENTS:
Time Frame: For the duration of the study (up to 2 years)
Arm/Group | Armodafinil 100 to 250 mg/Day
Serious Adverse Events (participants affected / at risk) | 56/731
Other Adverse Events (participants affected / at risk) | 667/731
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 100 to 250 mg/Day (N=731)
Myocardial infarction (Cardiac disorders) | 4
Coronary artery disease (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2
Abdominical adhesions (Gastrointestinal disorders) | 1
Abdominal Hernia (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Diverticulitis Intestinal (Gastrointestinal disorders) | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectocele (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 6
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 1
Choletithiasis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bursitis Infective (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pnuemonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Heat Stroke (Injury, poisoning and procedural complications) | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1
Cardioactive Drug Level Increased (Investigations) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Localised Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Intracranial Aneurysm (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 4
Cystocele (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Stress Incontinence (Renal and urinary disorders) | 1
Urethal Disorder (Renal and urinary disorders) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1
Uterine Polyp (Reproductive system and breast disorders) | 1
Uterine Prolapse (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Atherosclerosis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 100 to 250 mg/Day (N=731)
Nausea (Gastrointestinal disorders) | 68
Dry mouth (Gastrointestinal disorders) | 49
Diarrhoea (Gastrointestinal disorders) | 39
Nasopharyngitis (Infections and infestations) | 123
Upper respiratory tract infection (Infections and infestations) | 76
Sinusitis (Infections and infestations) | 64
Influenza (Infections and infestations) | 55
Bronchitis (Infections and infestations) | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 59
Back pain (Musculoskeletal and connective tissue disorders) | 53
Headache (Nervous system disorders) | 179
Dizziness (Nervous system disorders) | 47
Insomnia (Psychiatric disorders) | 99
Anxiety (Psychiatric disorders) | 57
Cough (Respiratory, thoracic and mediastinal disorders) | 42
Hypertension (Vascular disorders) | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days